CLINICAL TRIAL: NCT01156064
Title: Confocal Laser Endomicroscopy in Digestive Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Yang Yunsheng, Department of Gastroenterology and Hepatology
Other Study IDs: 07CX201
Record Dates: First submitted 2010-06-29; First posted 2010-07-02 (Estimated); Last update posted 2010-11-23 (Estimated); Status verified 2010-07

CONDITIONS: Digestive System Diseases
Keywords: Endoscopy; Confocal laser endomicroscopy; Digestive Diseases
MeSH Terms: conditions — Digestive System Diseases | interventions — Narrow Band Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — biopsy tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Case (subjects with digestive diseases): The investigators cases are subjects with confirmed digestive diseases.
  Interventions: Device: Confocal Laser Endomicroscopy (Pentax/Optiscan); Device: Narrow Band Imaging/Auto Fluorescence Imaging (Olympus)
- Control: Healthy individuals aged between 18 and 90 years who are asymptomatic for digestive diseases.
  Interventions: Device: Confocal Laser Endomicroscopy (Pentax/Optiscan); Device: Narrow Band Imaging/Auto Fluorescence Imaging (Olympus)

INTERVENTIONS:
Device: Confocal Laser Endomicroscopy (Pentax/Optiscan) — Confocal laser endomicroscopy is performed using the Pentax/Optiscan confocal endomicroscopy and 5 ml of 10% intravenous fluorescein sodium. Photos of magnified images of the digestive mucosa are taken during the procedure.
  Other Names: Confocal endomicroscopy
Device: Narrow Band Imaging/Auto Fluorescence Imaging (Olympus) — NBI/AFI endoscope offers an alternative light source involve NBI and AFI to view digestive mucosa in real time.
  Other Names: Narrow Band Imaging(NBI); Auto Fluorescence Imaging(AFI)

SUMMARY:
Confocal laser endomicroscopy (CLE) is a newly endoscopic device that enables microscopic view of the digestive tract. The purpose of this study is to determine if confocal laser endomicroscopy can improve detection of digestive disease include inflammation, dysplasia, and early cancer, and if confocal laser endomicroscopy has competitive advantage, compared with other device such as Narrow Band Imaging and Autofluoresecence Imaging.

DETAILED DESCRIPTION:
Advances in endoscopy have led to imagining of the details of digestive mucosa. Novel techniques such as Narrow Band Imaging (NBI) assisted magnification endoscopy, Auto Fluorescence Imaging (AFI) or confocal laser endomicroscopy could, however, improve the endoscopic detection.In this research we describe the combined use of these three techniques in patients with digestive disease.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over 18 years of age
* Subjects undergoing endoscopic procedures such as gastroscopy, colonoscopy, endoscopic retrograde cholangiopancreatography and endoscopic ultrasound will all be included

Exclusion Criteria:

* Under 18 years of age.
* Pregnancy or breast feeding
* Allergy to the fluorescent contrast agent fluorescein sodium
* Coagulopathy or bleeding disorder
* In emergency or life-threatening situations(eg. acute gastrointestinal hemorrhage, and gastrointestinal obstruction or perforation)
* impaired renal function, allergic asthma,
* Cognitively impaired.
* Residing in institutions (eg. prison, extended care facility)
* Have language barriers (eg. illiterate, dysphasic)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients of a tertiary referral hospital
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield for neoplasia of CLE vs. standard endoscopy | one year

SECONDARY OUTCOMES:
Diagnostic yield for neoplasia of CLE vs. NBI/AFI | one year

CONTACTS AND LOCATIONS:
Overall Officials: Yunsheng Yang, MD, Study Chair — Chinese PLA General Hospital
Locations (1):
- China PLA General Hospital, Beijing, Bejing, China

REFERENCES:
- [Derived] Huang J, Yang YS, Lu ZS, Wang SF, Yang J, Yuan J. Detection of superficial esophageal squamous cell neoplasia by chromoendoscopy-guided confocal laser endomicroscopy. World J Gastroenterol. 2015 Jun 14;21(22):6974-81. doi: 10.3748/wjg.v21.i22.6974. PMID 26078575